CLINICAL TRIAL: NCT03909529
Title: Two Way Crossover Oral Drug-drug Interaction Study of Spironolactone (Perpetrator) and Digoxin (Substrate Drug) in Healthy Adult Human Subjects Under Fasting Condition
Brief Title: Drug-drug Interaction (DDI) Study of Spironolactone (Perpetrator) and Digoxin (Substrate Drug)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CMP Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: C-CMP-SPI-001
Record Dates: First submitted 2019-02-16; First posted 2019-04-10 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-06

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — Digoxin; Tablets; Spironolactone

STUDY DESIGN:
Intervention Model Description: An open label, balanced, randomized, single-dose, two-treatment, two-sequence, two-period, crossover, drug-drug interaction study in healthy adult human subjects under fasting condition for spironolactone oral suspension (Carospir®)
Masking Description: Spironolactone Oral Suspension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LANOXIN® (Digoxin) USP 250 mcg (substrate drug) {Treatment A} (Experimental): 14 Subjects first administered with LANOXIN® (digoxin) USP 250 mcg (Substrate drug) on Day 6 of in house, after overnight fasting of at least 10.00 hours.
  After washout period of 28 days, these 14 subjects were administered with Spironolactone Oral Suspension 100 mg (perpetrator, Carospir® Oral Suspension 20 mL of 25 mg / 5 mL) from day 1 to day 5 and on day 6 the after overnight fasting of at least 10.00 hours, subject was administered with LANOXIN® (digoxin) USP 250 mcg (substrate drug) + Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL). From day 7 to day 9 the subjects were administered with Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL).
  Interventions: Drug: Digoxin 250 MCG Oral Tablet
- LANOXIN® (Digoxin) USP 250mcg and Carospir® Oral Suspension 20mL of 25 mg/5mL-Treatment B (Experimental): 14 Subjects first administered with Spironolactone Oral Suspension 100 mg (perpetrator, Carospir® Oral Suspension 20 mL of 25 mg / 5 mL) from day 1 to day 5 and on day 6 the after overnight fasting of at least 10.00 hours, subject was administered with LANOXIN® (digoxin) USP 250 mcg (substrate drug) + Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL). From day 7 to day 9 the subjects were administered with Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL).
  After washout period of 28 days these 14 Subjects administered with LANOXIN® (digoxin) USP 250 mcg (Substrate drug) on Day 6 of in house, after overnight fasting of at least 10.00 hours
  Interventions: Drug: Spironolactone 25 mg/ 5 mL S/F Suspension

INTERVENTIONS:
Drug: Digoxin 250 MCG Oral Tablet — The intervention is for study of drug drug interaction of digoxin when administered with spironolactone oral suspension
  Other Names: Spironolactone Oral Suspension 20 mL of 25 mg/mL
  Arms: LANOXIN® (Digoxin) USP 250 mcg (substrate drug) {Treatment A}
Drug: Spironolactone 25 mg/ 5 mL S/F Suspension — The intervention is for study of drug drug interaction of digoxin when administered with spironolactone oral suspension
  Other Names: DDI Spironolactone oral suspension interaction with digoxin
  Arms: LANOXIN® (Digoxin) USP 250mcg and Carospir® Oral Suspension 20mL of 25 mg/5mL-Treatment B

SUMMARY:
An open label, balanced, randomized, single-dose, two-treatment, two-sequence, two-period, crossover oral drug-drug interaction study of spironolactone (perpetrator) and Digoxin (substrate drug) in healthy adult human subjects under fasting condition.

DETAILED DESCRIPTION:
Drug interaction studies between spironolactone and digoxin, particularly studies in which digoxin was administered intravenously (Waldorf, S 1978; Fenster, P.E. 1984), indicate that spironolactone may decrease the renal clearance of digoxin by 18-25%, and increase the (area under curve) AUC of digoxin by 35-44%. Although the radioimmunoassay used in the study may be confounded, these results suggest that inhibition of P-gp in the renal proximal tubules may be possible. To account for possible renal P-gp inhibition, subjects in the test group will be pretreated with spironolactone for about 5 days to allow accumulation of some of the metabolites which have a long half-life (e.g., canrenone ~33 hours) and continue to be treated with spironolactone while digoxin is renally eliminated from the body. Based on this assessment, the FDA suggested study design is Treatment A: Single dose of digoxin alone. Treatment B: Digoxin + Spironolactone; Day 1- 9: Spironolactone single dose; Day 6: Digoxin single oral dose.

Also, digoxin has a long half-life of 1.5-2 days, and the Pharmacokinetic (PK) sampling scheme of up to 72 hours may not be enough to characterize the elimination kinetics of digoxin. Hence, the plasma concentrations of digoxin up to 96 hours (4 days) postdose is considered This will allow you to detect possible differences in the clearance of digoxin mediated by an interaction with P-gp in the renal proximal tubules.

The study also involves collecting urine samples and measuring renal clearance (CLR) and unchanged drug excreted in urine (fe) for digoxin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy human subjects aged between 20 and 35 years (including both).
* Subjects with a BMI between 18.5 - 24.9 Kg/m2 (including both) but body weight not less than 60 Kgs.
* Subjects who were screened at least 48 hours prior to check-in
* Subjects with normal health as determined by personal medical history, clinical examination, and laboratory examinations including serological tests during the screening
* Subjects with normal 2D echo
* Subjects having normal 12-lead electrocardiogram (ECG) or ECG with no clinical significant abnormalities as determined by Investigator.
* Subjects having normal chest X-Ray (P/A view) or chest X-ray with no clinically significant abnormalities as determined by investigator.
* Subjects able to communicate effectively.
* Subjects willing to give written informed consent and adhere to all the requirements of this protocol.
* Additional inclusion criteria for female subjects, Female of childbearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence: or Postmenopausal for at least 1 year, or Surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed on the subject).

Exclusion Criteria:

* Subjects having contraindications or hypersensitivity to study drug or related group of drugs.
* History or presence of any medical condition or disease according to the opinion of the physician.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
* Subject having QT/ corrected QT interval (QTc) >450 milliseconds
* History or presence of significant alcoholism or drug abuse in the past one year.
* History or presence of significant smoking (more than 10 cigarettes /day or consumption of tobacco products).
* Subjects who fail to abstain from consuming any alcoholic products from 48.00 hours prior to check-in to till check-out / last sample of the study.
* Subjects who fail to abstain from any xanthine-containing food and/or beverages (like chocolate, tea, coffee, cola drinks), cigarettes and tobacco containing products and grapefruit and/or it's juice from 48.00 hours prior to check-in to till check-out / last sample of the study.
* Subjects who fail to refrain from pan or pan masala, gutkha, masala (containing beetle nut and tobacco) for 48.00 hours prior to check-in to till check-out/last sample of the study.
* Difficulty with donating blood.
* Systolic blood pressure less than 110 mm Hg or more than 140 mm Hg.
* Diastolic blood pressure less than 70 mm Hg or more than 90 mm Hg.
* Pulse rate less than 60 beats/minute or more than 100 beats/minute.
* Use of any prescribed medication during last two weeks or over-the- counter (OTC) medicinal products/ herbal products during the last one week prior to check-in.
* Major illness during 90 days before check-in.
* Participation in a drug research study within past 90 days of check-in.
* Donation of blood (i.e. one unit or 350 mL) in the past 90 days before check-in.
* History of unusual diet consumption in the past 3 weeks before check-in.
* Additional exclusion criteria for female subjects, Volunteer demonstrating a positive pregnancy test. Volunteers who are pregnant, currently breast-feeding or who are likely to become pregnant during the study.

Volunteers who have used implanted or injected hormonal contraceptives anytime during the 6 months prior to study or used hormonal contraceptives within 14 days before dosing.

-

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopali K Somani, MD, Principal Investigator — Employee
Locations (1):
- ClinSync Clinical Research Pvt. Ltd., Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- LANOXIN First, Then Carospir: 14 Subjects first administered with LANOXIN® (digoxin) USP 250 mcg (Substrate drug) on Day 6 of in house, after overnight fasting of at least 10.00 hours.
  After washout period of 28 days, these 14 subjects were administered with Spironolactone Oral Suspension 100 mg (perpetrator, Carospir® Oral Suspension 20 mL of 25 mg / 5 mL) from day 1 to day 5 and on day 6 the after overnight fasting of at least 10.00 hours, subject was administered with LANOXIN® (digoxin) USP 250 mcg (substrate drug) + Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL). From day 7 to day 9 the subjects were administered with Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL)
- First Carospir, Then LANOXIN: 14 Subjects first administered with Spironolactone Oral Suspension 100 mg (perpetrator, Carospir® Oral Suspension 20 mL of 25 mg / 5 mL) from day 1 to day 5 and on day 6 the after overnight fasting of at least 10.00 hours, subject was administered with LANOXIN® (digoxin) USP 250 mcg (substrate drug) + Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL). From day 7 to day 9 the subjects were administered with Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL).
  After washout period of 28 days these 14 Subjects administered with LANOXIN® (digoxin) USP 250 mcg (Substrate drug) on Day 6 of in house, after overnight fasting of at least 10.00 hours
Period: Open Label, Balanced, Randomized DDI
Arm/Group | LANOXIN First, Then Carospir | First Carospir, Then LANOXIN
Started | 14 (14 Subjects received this treatment) | 14 (14 Subjects received this treatment)
Completed | 14 (14 subjects completed this treatment) | 14 (14 Subjects completed this treatment)
Not Completed | 0 | 0
Period: Open Label, Balanced, Randomized DDI
Arm/Group | LANOXIN First, Then Carospir | First Carospir, Then LANOXIN
Started | 14 (14 Subjects received this treatment) | 14 (14 Subjects received this treatment)
Completed | 14 (14 subjects completed this treatment) | 14 (14 subjects completed this treatment)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: On Day 6 of each period, after overnight fasting for at least 10.00 hours the subjects were dosed either with the Treatment (A) [LANOXIN® (digoxin) USP 250 mcg (substrate drug)] or Treatment (B) [LANOXIN® (digoxin) USP 250 mcg (substrate drug) + Spironolactone Oral Suspension 100 mg (Perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL)] as per the randomization scheme.
Groups:
- Drug-Drug Interaction Study: In both periods (Period-I and II), from Day 1 to Day 5 and Day 7 to Day 9, the subjects who were randomized to treatment B, were administered Spironolactone Oral Suspension 100 mg (Perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL), and the subject who were randomized to treatment A were not dosed.
  On all these days the standard breakfast was served 0.50 hr (30 min) post dose.
  On Day 6, after overnight fasting for at least 10.00 hours the subjects were dosed either with the Treatment (A) [LANOXIN® (digoxin) USP 250 mcg (substrate drug)] or Treatment (B) [LANOXIN® (digoxin) USP 250 mcg (substrate drug) + Spironolactone Oral Suspension 100 mg (Perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL)] as per the randomization scheme.
Arm/Group | Drug-Drug Interaction Study
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 29 [23 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  India | 28

OUTCOME MEASURES:

1. Primary Outcome: Dogoxin Plasma Data for Cmax
Description: Primary Pharmacokinetic parameter The following pharmacokinetic parameters for Digoxin were obtained using non-compartmental method Cmax, AUC0-96, and tmax using plasma data, Renal clearance (CLR) /Percent Recovered, Unchanged drug excreted in urine (fe)/Amount Recovered using urine data.
Time Frame: 4 days
Population: The following pharmacokinetic parameters for Digoxin were obtained using non-compartmental method (WinNonlin, version 8.1, Pharsight Corporation, USA):
  Cmax, AUC0-96, and tmax using plasma data, Renal clearance (CLR) /Percent Recovered, Unchanged drug excreted in urine (fe)/Amount Recovered using urine data.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Drug-Drug Interaction Study: This was an open label, balanced, randomized, single-dose, two-treatment, two-sequence, two-period, crossover, drug drug interaction study in healthy adult human subjects with at least 28 days washout period between each treatment period under fasting condition
  In both periods (Period-I and II), from Day 1 to Day 5 and Day 7 to Day 9, the subjects who were randomized to treatment B, were administered Spironolactone Oral Suspension 100 mg (Perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL), and the subject who were randomized to treatment A were not dosed.
  On Day 6, after overnight fasting for at least 10.00 hours the subjects were dosed either with the Treatment (A) [LANOXIN® (digoxin) USP 250 mcg (substrate drug)] or Treatment (B) [LANOXIN® (digoxin) USP 250 mcg (substrate drug) + Spironolactone Oral Suspension 100 mg (Perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL)] as per the randomization scheme.
Arm/Group | Drug-Drug Interaction Study
Number analyzed (Participants) | 28
pg/mL
  Treatment A | 1530.188 (502.810)
  Treatment B | 2432.908 (870.562)

2. Primary Outcome: Digoxin Plasma Data for AUC0-96
Description: Area under the plasma concentration versus time curve from time 0 to the 96 hour time point concentration.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: pg.hr/mL
Groups:
- Drug-Drug Interaction Study: In both periods (Period-I and II), from Day 1 to Day 5 and Day 7 to Day 9, the subjects who were randomized to treatment B, were administered Spironolactone Oral Suspension 100 mg (Perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL), and the subject who were randomized to treatment A were not dosed.
  On Day 6, after overnight fasting for at least 10.00 hours the subjects were dosed either with the Treatment (A) [LANOXIN® (digoxin) USP 250 mcg (substrate drug)] or Treatment (B) [LANOXIN® (digoxin) USP 250 mcg (substrate drug) + Spironolactone Oral Suspension 100 mg (Perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL)] as per the randomization scheme.
Arm/Group | Drug-Drug Interaction Study
Number analyzed (Participants) | 28
pg.hr/mL
  Treatment A | 13715.974 (2669.003)
  Treatment B | 16551.500 (4108.500)

3. Secondary Outcome: Digoxin Plasma Data for Tmax
Description: If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value.
Time Frame: 4 days
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Drug-Drug Interaction Study
Number analyzed (Participants) | 28
hr
  Treatment A | 0.744 (0.195)
  Treatment B | 0.901 (0.569)

4. Secondary Outcome: ECG Measurement Will be Performed to Evaluate Any Changes in the QT Interval
Description: ECG will be performed at 1.00 and 3.00 hours post dose in each period on Day 6 and at check-out of each period of the study
Time Frame: 4 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Renal Clearance (CLR)/Percent Recovered
Description: Summary Statistics for Untransformed Urine PK Parameters of digoxin Per Treatment-Renal clearance (CLR)/Percent Recovered
Time Frame: 04 Days
Measure: Mean (Standard Deviation); unit: % recovered
Arm/Group | Drug-Drug Interaction Study
Number analyzed (Participants) | 28
% recovered
  Treatment A | 54.687 (29.158)
  Treatment B | 53.378 (21.256)

6. Other Pre Specified Outcome: Unchanged Drug Excreted in Urine (fe)/ Amount Recovered
Description: Summary of Urine Pharmacokinetic parameters for digoxin -unchanged drug excreted in urine (fe)/ Amount Recovered
Time Frame: 04 Days
Measure: Mean (Standard Deviation); unit: nanograms
Arm/Group | Drug-Drug Interaction Study
Number analyzed (Participants) | 28
nanograms
  Treatment A | 136717.72 (72895.492)
  Treatment B | 133446.07 (53141.044)

ADVERSE EVENTS:
Time Frame: 9 days for period 18 Days for 2 periods
Groups:
- Treatment-A- Single Dose of Digoxin (LANOXIN): 14 Subjects first administered with LANOXIN® (digoxin) USP 250 mcg (Substrate drug) on Day 6 of in house, after overnight fasting of at least 10.00 hours in period I.
  After washout period of 28 days, in period II another 14 subjects (other than first 14 subjects) were administered with LANOXIN® (digoxin) USP 250 mcg (Substrate drug) on day 6 the after overnight fasting of at least 10.00 hours.
- Treatment-B-Digoxin (LANOXIN) + Spiranolactone (Carospir): 14 Subjects first administered with Spironolactone Oral Suspension 100 mg (perpetrator, Carospir® Oral Suspension 20 mL of 25 mg / 5 mL) from day 1 to day 5 and on day 6 the after overnight fasting of at least 10.00 hours in period I. From day 7 to day 9 the subjects were administered with Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL).
  After washout period of 28 days, in period II another 14 subjects (other than first 14 subjects) were administered with Spironolactone Oral Suspension 100 mg (perpetrator, Carospir® Oral Suspension 20 mL of 25 mg / 5 mL) from day 1 to day 5 and on day 6 the after overnight fasting of at least 10.00 hours. From day 7 to day 9 the subjects were administered with Spironolactone Oral Suspension 100 mg (perpetrator; Carospir® Oral Suspension 20 mL of 25 mg / 5 mL).
Arm/Group | Treatment-A- Single Dose of Digoxin (LANOXIN) | Treatment-B-Digoxin (LANOXIN) + Spiranolactone (Carospir)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03909529/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03909529/SAP_001.pdf